CLINICAL TRIAL: NCT00177320
Title: Rheumatic Diseases and Computer Use: A Needs Assessment
Brief Title: Rheumatic Diseases and Computer Use
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Nancy Baker, Nancy A. Baker, University of Pittsburgh
Other Study IDs: 0502148
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2016-01-25 (Estimated); Status verified 2016-01

CONDITIONS: Rheumatoid Arthritis; Fibromyalgia; Osteoarthritis
Keywords: Rheumatic Disorders; Computer Use
MeSH Terms: conditions — Arthritis, Rheumatoid; Fibromyalgia; Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Computers allow individuals to engage in economic, social, and entertainment activities. Despite the many benefits of computer use, many individuals with rheumatic diseases may have difficulty using a computer. However, currently there is almost no information on the problems individuals with rheumatic diseases experience using a computer. Baseline information on the types of problems experienced by individuals with rheumatic diseases as well as the magnitude of those problems is needed before methods can be developed to intervene and remediate them. In this study we will develop and administer to a representative sample of patients with rheumatic diseases a survey which will examine the type and magnitude of computer problems experienced by those with rheumatic diseases. The goal of this study is to complete a needs assessment on the problems experienced by those with rheumatic diseases during computer use. This assessment will lay the groundwork for the development of outcome measures and interventions to improve computer use for individuals with rheumatic diseases. In the future it will assist individuals with rheumatic diseases to be able to use computers more comfortably and efficiently.

DETAILED DESCRIPTION:
Computers allow individuals to engage in economic, social, and entertainment activities. They are vital for full participation in many areas of society, and have become a necessity for many types of employment, particularly management and administrative positions. Despite the many benefits of computer use, many individuals with rheumatic diseases such as rheumatoid arthritis (RA), osteoarthritis (OA), and fibromyalgia (FM) may be unable to use a computer due to limitations in hand function or sitting ability. These limitations can prevent the physical manipulation of computer peripherals or inhibit the ability to sit for extended periods of time at a computer. Despite the importance of computer use there is almost no information on the problems individuals with rheumatic diseases experience using a computer. Baseline information on the types of problems experienced by individuals with rheumatic diseases as well as the magnitude of those problems is needed before methods can be developed to intervene and remediate them. The aim of this study is to complete a needs assessment on the problems experienced by those with rheumatic diseases during computer use. This assessment will lay the groundwork for the development of outcome measures and interventions to improve computer use for individuals with rheumatic diseases by identifying problem areas and examine the magnitude of those problems. This study will be implemented in two phases. In Phase I (months 01-05) we will use several focus group sessions of 5-10 participants to acquire consumer input to develop and refine a survey to examine the problems experienced during computer use by people with rheumatic diseases. In Phase II the survey developed in Phase I {Computer Problem Survey (ComPS)] will be administered to a representative sample of patients with rheumatic diseases (n = ~1500) to ascertain the type and magnitude of computer problems (months 06-12). These 2 phases will be used to answer the following questions: 1. What aspects of computer use are reported to be a problem for individuals with RA, OA, and FM? 2. What is the magnitude of these problems for individuals with RA, OA, and FM? 3. How does the magnitude differ when examined by age, gender, education, race/ethnicity, and work status? At the end of the study we will have gathered the descriptive data necessary to 1) begin modifying current computer performance evaluations to focus on measuring computer use performance in individuals with rheumatic diseases; and 2) develop and test interventions, such as adaptive equipment and ergonomics, to promote continued computer use for individuals with difficulties using a computer due to physical limitations.

ELIGIBILITY:
Inclusion Criteria:

* Has Fibromyalgia, Osteoarthritis, or Rheumatoid arthritis; between 18-65; in the UPMC Arthritis Network Disease REgistry

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Respondents were recruited from the University of Pittsburgh Medical Center Arthritis Network Disease Registry,
Sampling Method: Non-Probability Sample
Enrollment: 359 (Actual)
Dates: Start 2005-03; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy A. Baker, ScD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States